CLINICAL TRIAL: NCT00466635
Title: An Open-label Study to Assess the Safety, Efficacy and Absorption of Exodif™ (Tolevamer Potassium Sodium) Tablets in Patients With Clostridium Difficile-Associated Diarrhea
Brief Title: A Study to Assess the Safety, Tolerability, Effectiveness and Absorption of Exodif™ Tablets in Clostridium Difficile-associated Diarrhea
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOL26700706
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Enterocolitis, Pseudomembranous; Diarrhea; Clostridium Difficile
Keywords: Clostridium difficile Disease; Infectious diarrhea; C. difficile; CDAD; Clostridium difficile-associated diarrhea; Clostridium difficile diarrhea; Antibiotic-Associated Colitis; Clostridium Enterocolitis; Antibiotic-Associated Diarrhea; Pseudomembranous Colitis; Clostridium difficile
MeSH Terms: conditions — Enterocolitis, Pseudomembranous; Diarrhea; Dysentery

INTERVENTIONS:
Drug: GT267-004 (tolevamer potassium sodium)

SUMMARY:
Approximately 65 patients will be entered into this study taking place in North America. The aim of this study is to evaluate the safety, efficacy and absorption of an investigational drug in patients with C. difficile-associated diarrhea (CDAD). All study related care is provided including doctor visits, physical exams, laboratory tests and study medication. Total length of participation is 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The presence of CDAD at the time of enrollment
* Negative serum pregnancy test (HCG) for women of childbearing potential.

Exclusion Criteria:

* Any contraindication to oral / enteral therapy including fulminant C. difficile disease.
* Any acutely life-threatening medical conditions.
* Acute or chronic diarrhea of other cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2007-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Clinical Success
Safety

SECONDARY OUTCOMES:
The extent of tolevamer absorption

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (13):
- United States (13):
  - Modesto, California
  - Honolulu, Hawaii
  - Maywood, Illinois
  - Baltimore, Maryland
  - Worcester, Massachusetts
  - West Bloomfield, Michigan
  - Butte, Montana
  - Cedar Knolls, New Jersey
  - Neptune City, New Jersey
  - Syracuse, New York
  - Greenville, North Carolina
  - Toledo, Ohio
  - Lancaster, Pennsylvania